CLINICAL TRIAL: NCT00975507
Title: A Pilot Study to Compare the Safety, Tolerability, and Immunogenicity of Measles, Mumps, Rubella, and Varicella (MMRV) Vaccine and the Concomitant Administration of the Currently Licensed VARIVAX™ and M-M-R II™ in Healthy Children
Brief Title: ProQuad™ Versus M-M-R II™ and VARIVAX™ in Healthy Children (V221-009)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V221-009; 2009_660
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ProQuad™ (V221) + Placebo Followed by ProQuad™
  Interventions: Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live; Biological: Comparator: Placebo
- 2 (Active Comparator): M-M-R™ II + VARIVAX™
  Interventions: Biological: Comparator: Varivax; Biological: Comparator: M-M-R II

INTERVENTIONS:
Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live — a single 0.5 mL subcutaneous injection of V221 at Day 0 and Day 90
  Other Names: ProQuad™
  Arms: 1
Biological: Comparator: Placebo — a single 0.5 mL subcutaneous placebo injection at Day 0
  Arms: 1
Biological: Comparator: Varivax — a single 0.5 mL subcutaneous injection of Varivax at Day 0
  Arms: 2
Biological: Comparator: M-M-R II — a single 0.5 mL subcutaneous injection of M-M-R II at Day 0
  Arms: 2

SUMMARY:
This study will compare Measles, Mumps, Rubella, and Varicella Vaccine (V221) and concomitant administration of Varivax and M-M-R II vaccines in healthy children.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* Negative clinical history of varicella, shingles, measles, mumps, and rubella

Exclusion Criteria:

* Previous receipt of measles, mumps, rubella and/or varicella vaccine either alone or in combination
* Any immune impairment or deficiency
* Exposure to measles, mumps, rubella, varicella, or zoster in the 4 weeks prior to vaccination
* Vaccination with an inactive vaccine with in the past 14 days
* Vaccination with a live vaccine within the past 30 days
* Immune globulin or any blood product administered in the past 3 months

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 1998-03; Primary Completion 1999-01 (Actual); Study Completion 1999-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Shinefield H, Black S, Digilio L, Reisinger K, Blatter M, Gress JO, Brown ML, Eves KA, Klopfer SO, Schodel F, Kuter BJ. Evaluation of a quadrivalent measles, mumps, rubella and varicella vaccine in healthy children. Pediatr Infect Dis J. 2005 Aug;24(8):665-9. doi: 10.1097/01.inf.0000172902.25009.a1. PMID 16094217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 clinical sites in the United States
  Date of first participant visit: 24-Mar-1998
  Date of last participant visit: 05-Jan-1999
Groups:
- ProQuad™ + Placebo Followed by ProQuad™: ProQuad™ (measles, mumps, rubella, and varicella vaccine) containing a high varicella component (~40,000 PFU/0.5 mL-dose) with a standard measles component (~3.7 log10 TCID50/0.5 mL dose) + placebo administered concomitantly at separate injection sites on Day 0. Second dose of ProQuad™ containing a high varicella component (~40,000 PFU/0.5 mL-dose) with a standard measles component (~3.7 log10 TCID50/0.5 mL dose) administered approximately 90 days (Day 90) after the first dose.
- M-M-R™ II + VARIVAX™: VARIVAX™ + M-M-R™ II administered concomitantly at separate injection sites on Day 0.
Period: Overall Study
Arm/Group | ProQuad™ + Placebo Followed by ProQuad™ | M-M-R™ II + VARIVAX™
Started | 323 | 157
Vaccinated at Visit 1 | 323 | 157
Vaccinated at Visit 2 | 310 | 0 (Per-protocol, subjects receiving M-M-R™ II + VARIVAX™ at Visit 1 were not vaccinated at Visit 2)
Completed | 303 | 153
Not Completed | 20 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 7 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 10 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ProQuad™ + Placebo Followed by ProQuad™ | M-M-R™ II + VARIVAX™ | Total
Number analyzed (Participants) | 323 | 157 | 480
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.1 (1.9) | 14.0 (1.7) | 14.1 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 87 | 260
  Male | 150 | 70 | 220
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 41 | 21 | 62
  Asian/Pacific | 30 | 9 | 39
  Caucasian | 211 | 107 | 318
  Hispanic | 30 | 16 | 46
  Other | 11 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postvaccination Varicella Antibody Titer ≥5 Glycoprotein Enzyme-Linked Immunosorbent Assay (gpELISA) Units/mL for Subjects Initially Seronegative (a Titer of <0.6 gpELISA Units/mL) to Varicella at Baseline
Description: Antibody Response to Varicella at 6 Weeks Postvaccination for Subjects Initially Seronegative (a titer of <0.6 gpELISA units/mL) to Varicella at Baseline
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to varicella at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™+Placebo Followed by ProQuad™ - (1 Injection ProQuad™) | ProQuad™+Placebo Followed by ProQuad™ - (2 Injection ProQuad™) | M-M-R™ II + VARIVAX™ (1 Injection)
Number analyzed (Participants) | 250 | 239 | 128
Participants | 228 | 237 | 118

2. Secondary Outcome: Number of Participants With Postvaccination Measles ELISA Antibody Titer ≥207.8 mIU/mL
Description: Antibody Response to Measles at 6 Weeks Postvaccination for Subjects Initially Seronegative (a titer <207.8 mIU/mL) to Measles at Baseline
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to measles at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™+Placebo Followed by ProQuad™ - (1 Injection ProQuad™) | ProQuad™+Placebo Followed by ProQuad™ - (2 Injection ProQuad™) | M-M-R™ II + VARIVAX™ (1 Injection)
Number analyzed (Participants) | 302 | 288 | 145
Participants | 290 | 284 | 145

3. Secondary Outcome: Number of Participants With Postvaccination Varicella Antibody Titer ≥5 gpELISA Units/mL for Subjects Initially With Varicella Antibody Titer <1.25 gpELISA Units/mL at Baseline
Description: Antibody Response to Varicella at 6 Weeks Postvaccination for Subjects Initially With Varicella Antibody Titer <1.25 gpELISA units/mL at Baseline
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, Varicella Antibody Titer <1.25 gpELISA units/mL at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™+Placebo Followed by ProQuad™ - (1 Injection ProQuad™) | ProQuad™+Placebo Followed by ProQuad™ - (2 Injection ProQuad™) | M-M-R™ II + VARIVAX™ (1 Injection)
Number analyzed (Participants) | 290 | 278 | 145
Participants | 264 | 275 | 134

4. Secondary Outcome: Number of Participants With Postvaccination Mumps ELISA Antibody Titer ≥2.0 Ab Units/mL
Description: Antibody Response to Mumps at 6 Weeks Postvaccination for Subjects Initially Seronegative (a titer <2.0 Ab Units/mL) to Mumps at Baseline
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to mumps at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™+Placebo Followed by ProQuad™ - (1 Injection ProQuad™) | ProQuad™+Placebo Followed by ProQuad™ - (2 Injection ProQuad™) | M-M-R™ II + VARIVAX™ (1 Injection)
Number analyzed (Participants) | 295 | 283 | 150
Participants | 292 | 283 | 148

5. Secondary Outcome: Number of Participants With Postvaccination Rubella ELISA Antibody Titer ≥10 IU/mL
Description: Antibody Response to Rubella at 6 Weeks Postvaccination for Subjects Initially Seronegative (a titer <10 IU/mL) to Rubella at Baseline
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to rubella at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™+Placebo Followed by ProQuad™ - (1 Injection ProQuad™) | ProQuad™+Placebo Followed by ProQuad™ - (2 Injection ProQuad™) | M-M-R™ II + VARIVAX™ (1 Injection)
Number analyzed (Participants) | 304 | 290 | 153
Participants | 289 | 275 | 142

ADVERSE EVENTS:
Description: The number of participants listed as "at risk" is the number of participants with follow-up.
Groups:
- ProQuad™ + Placebo Then ProQuad™ - ProQuad™ (1 Injection): ProQuad™ (measles, mumps, rubella, and varicella vaccine) containing a high varicella component (~40,000 PFU/0.5 mL-dose) with a standard measles component (~3.7 log10 TCID50/0.5 mL dose) + placebo administered concomitantly at separate injection sites on Day 0.
- ProQuad™ + Placebo Then ProQuad™ - ProQuad™ (2 Injections): ProQuad™ (measles, mumps, rubella, and varicella vaccine) containing a high varicella component (~40,000 PFU/0.5 mL-dose) with a standard measles component (~3.7 log10 TCID50/0.5 mL dose) + placebo administered concomitantly at separate injection sites on Day 0. Second dose of ProQuad™ containing a high varicella component (~40,000 PFU/0.5 mL-dose) with a standard measles component (~3.7 log10 TCID50/0.5 mL dose) administered approximately 90 days (Day 90) after the first dose.
- M-M-R™ II + VARIVAX™ (1 Injection): VARIVAX™ + M-M-R™ II administered concomitantly at separate injection sites on Day 0.
Arm/Group | ProQuad™ + Placebo Then ProQuad™ - ProQuad™ (1 Injection) | ProQuad™ + Placebo Then ProQuad™ - ProQuad™ (2 Injections) | M-M-R™ II + VARIVAX™ (1 Injection)
Serious Adverse Events (participants affected / at risk) | 0/321 | 1/308 | 1/156
Other Adverse Events (participants affected / at risk) | 238/321 | 190/308 | 110/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ProQuad™ + Placebo Then ProQuad™ - ProQuad™ (1 Injection) (N=321) | ProQuad™ + Placebo Then ProQuad™ - ProQuad™ (2 Injections) (N=308) | M-M-R™ II + VARIVAX™ (1 Injection) (N=156)
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 1
Infection, rotovirus (Infections and infestations) | 0 | 0 | 1
Infection, viral (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ProQuad™ + Placebo Then ProQuad™ - ProQuad™ (1 Injection) (N=321) | ProQuad™ + Placebo Then ProQuad™ - ProQuad™ (2 Injections) (N=308) | M-M-R™ II + VARIVAX™ (1 Injection) (N=156)
Fever (General disorders) | 129 | 72 | 54
Infection, Viral (Infections and infestations) | 8 | 6 | 7
Trauma (Injury, poisoning and procedural complications) | 1 | 4 | 3
Hemorrhage, Venipuncture Site (Injury, poisoning and procedural complications) | 0 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 14 | 8 | 1
Diarrhea (Gastrointestinal disorders) | 29 | 19 | 13
Gastroenteritis (Gastrointestinal disorders) | 4 | 3 | 2
Gastroenteritis, Infectious (Infections and infestations) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 3
Teething (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 18 | 5 | 12
Headache (Nervous system disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 6 | 3 | 3
Irritability (Psychiatric disorders) | 39 | 23 | 16
Somnolence (Psychiatric disorders) | 4 | 2 | 3
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Congestion, Nasal (Respiratory, thoracic and mediastinal disorders) | 1 | 11 | 2
Congestion, Respiratory (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 25 | 6
Infection, Respiratory, Upper (Infections and infestations) | 34 | 73 | 11
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 2
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 18 | 18 | 8
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0
Bite/Sting, Non-Venomous (Injury, poisoning and procedural complications) | 6 | 1 | 2
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 2
Dermatitis, Contact (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Dermatomycosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 7 | 2 | 0
Miliaria Rubra (Skin and subcutaneous tissue disorders) | 9 | 1 | 8
Rash (Skin and subcutaneous tissue disorders) | 29 | 13 | 16
Rash, Measles/Rubella-Like (Skin and subcutaneous tissue disorders) | 18 | 4 | 3
Rash, Varicella-Like (Skin and subcutaneous tissue disorders) | 7 | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 6 | 5 | 2
Viral Exanthema (Skin and subcutaneous tissue disorders) | 17 | 4 | 9
Conjunctivitis (Eye disorders) | 4 | 5 | 1
Otitis (Ear and labyrinth disorders) | 7 | 1 | 3
Otitis (Ear and labyrinth disorders) | 19 | 13 | 4
Erythema (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 9 | 7 | 0/0
Pain/Tenderness/Soreness (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 9 | 9 | 0/0
Rash (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 5 | 0 | 0/0
Swelling (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 6 | 3 | 0/0
Ecchymosis (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 5
Erythema (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 8
Pain/Tenderness/Soreness (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 3
Swelling (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 2
Pain/Tenderness/Soreness (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.